CLINICAL TRIAL: NCT06081010
Title: Community Health Worker Led Hypertension Prevention and Control (CHPC) in Nepal: An Implementation Trial
Brief Title: FCHV-HTN Implementation Trial in Nepal
Acronym: CHPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Dhulikhel Hospital (Other); Institute for Implementation Science and Health (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000036053; 1R01HL169421-01 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
Keywords: Hypertension; Community Health Worker; Implementation Trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Community Health Worker Intervention
  Interventions: Behavioral: Community Health Worker Intervention
- Control Group (No Intervention): Usual care that includes patients visit to health facility based on felt need

INTERVENTIONS:
Behavioral: Community Health Worker Intervention — Trained CHWs will hold group meetings or home visits using a locally adapted manual for HTN management. CHWs will visit homes in their areas and measure BP. High BP clients will be taken to the nearest health center. CHWs will enroll individuals with preHTN and HTN and conduct 4 follow-up group meetings or home visits with them every 3 months. Participants will be invited to attend CHW lead group-based counseling. For those with uncontrolled HTN who have difficulty adhering to prescribed HTN management and not willing or able to attend group meetings, CHWs will conduct follow-up home visits. First meeting (about 90 minutes), CHWs will explain purpose of the meeting and discuss HTN and its consequences. CHWs will apply techniques to initiate dialogue and reflection regarding lifestyle modifications and choose goals based on PEN protocol-2, BP monitoring, and antihypertensive medication use. In subsequent meetings (about 60 minutes), the CHWs will measure BP and address ongoing problems.
  Arms: Intervention arm

SUMMARY:
The goal of this hybrid type III study incorporating a cluster-randomized trial is to assess the effect of a community health worker-led hypertension prevention and control program (CHPC) on the implementation outcomes and clinical outcomes among patient with hypertension in central Nepal. The main questions it aims to answer are:

1. What is the level of implementation outcomes, including reach, adoption, implementation fidelity, and maintenance of the CHPC implementation strategy at the patient, provider, and health system levels?

2: What is the effectiveness of the CHPC implementation strategy compared to facility-based intervention on systolic BP via a cluster randomized controlled trial.

3: What is the implementation cost and cost-effectiveness of the CHPC implementation strategy?

Participants will receive four follow-up group meetings or home visits every three months for a year by a community health worker. Researchers will compare if there is a significant difference in systolic blood pressure between those who receive this intervention and those who do not receive the intervention in the same community.

DETAILED DESCRIPTION:
INTRODUCTION:

Hypertension (HTN) is a global public health challenge. About 13.5% of global total mortality is attributed to high blood pressure (BP) worldwide. In addition, about 54% of strokes and 47% of coronary heart disease worldwide were attributable to high BP. In Nepal, the adult HTN prevalence is 25%, similar to the global prevalence. Community Health Workers (CHWs) are the frontline pillars of community-based health programs in Nepal. Through CHW, this investigation aims to influence HTN control and behavior change among adults and society at large. By providing a replicable model for increasing HTN awareness, treatment, and control in Nepal, investigators will accelerate the integration of effective intervention into practice, providing an example of amelioration of the well-documented delays in moving tested interventions to practice. To ensure relevance to policymakers, the investigators will follow the principles of 'practical trials that include: (a) implementing the strategy, (b) facilitating and evaluating the maintenance of the strategy beyond the implementation phase; (c) using multiple evaluation measures relevant to decision makers, including reach, adoption, and cost; and (d) evaluating effectiveness across multiple outcomes, with a plan to triangulate findings from across multiple data sources using both qualitative and quantitative measures.

METHODS:

Investigators will conduct a Hybrid type III effectiveness-implementation design focusing primarily on implementation outcomes while also collecting effectiveness outcomes as they relate to the uptake or fidelity of the intervention. The primary implementation outcomes (aim 1) - reach, adoption, implementation and maintenance - are selected to answer the central research question of this study and will be assessed using a non-inferiority design. Investigators will assess these outcomes in the intervention group using data from the process evaluation in intervention health facilities. For each outcome, the null hypothesis is that the percentages are equivalent to a set target or greater. Thus, if the program is successful, investigators will be able to say with 95% confidence that these high standards have been met. To measure the effectiveness (aim 2), investigators will use a cluster-randomized design to assess change in mean systolic BP in the intervention group compared to the control group at 12 months after the intervention. Investigators will also measure cost and estimate incremental cost per participant with awareness on and control of high BP (aim 3).

STUDY SETTING:

We will conduct the study in Sindhupalchowk district, one of the largest districts in Bagmati province, Nepal, consisting of nine rural and three urban municipalities. Basic health facilities in the Sindhupalchowk district province that host CHWs will be included. In the study districts, there are 102 basic health facilities, and approximately 687 CHWs. These CHWs are female community health volunteers (FCHV) who provide basic health services in Nepal, historically focused on maternal and child health.

INTERVENTION: FCHV-led Hypertension Prevention and Control (CHPC) Program

Fundamentally, the intervention involves task-shifting of HTN management roles to primary care and community-level health workers, integrating the five components of the evidence-based interventions outlined in the Package of Essential Non-Communicable Diseases (PEN) protocol 1 and 2:

1. BP measurement and monitoring;
2. identify high BP individuals and report to health facility;
3. provide one-on-one counseling and lifestyle modification goal setting including sodium reduction, healthy diet, alcohol abstinence, physical activity, and medication;
4. BP monitoring of HTN patients; and
5. medication adherence of HTN patients, delivered by the FCHVs trained for the intervention.

The intervention will be conducted over a fiscal year, and repeated during the maintenance.

IMPLEMENTATION STRATEGIES:

To address barriers of implementing the intervention, we will incorporate the following strategies and core components:

1. Leadership support and ongoing program promotion - Health Coordinators from Provincial MoH will participate in the planning, execution and monitoring of the study. In provincial MoH health review meetings, hypertension-related indicators (proportion of population screened, HTN detected, HTN under medication, HTN control) will be discussed using the government's health management information system data.
2. Capacity building - Healthcare workers training; FCHV training; Coaching and technical support from healthcare workers to FCHV in a monthly meeting
3. CHW home visit and group meeting - 1st visit: introduction, rapport building, goal setting, BP monitoring; 2nd- 4th visit: BP monitoring, action and reflection, discussing problems faced in achieving their goals and implementing their action plans
4. Social network - Monthly meeting of health care workers in the municipality; Monthly meeting of FCHVs in the health facility

DATA SOURCES:

Quantitative - Participant Survey; Anthropometric Measurement; Blood Pressure Measurement; Healthcare Provider Survey; Process Tracking

Qualitative - Periodic Reflection; Meeting Observations; Focus Group Discussions; Key Informant Interviews

The primary aim is to determine the extent to which this implementation model meets acceptable rates of program adoption, implementation, reach and maintenance of the CHPC program. For assessing the adoption, implementation, reach, and maintenance, we will include all intervention health facilities. To assess the effectiveness, we are planning for patients to be enrolled over six months.

ELIGIBILITY:
Inclusion Criteria:

-High blood pressure (BP) of 140/90 mmHg or higher.

Exclusion Criteria:

* Severe illness requiring bed rest
* Pregnant women, due to their special health needs

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3572 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach | 12 months
  Percentage of CHWs implementing the program
Adoption | 12 months
  Percentage of the health facilities asked to participate in adopting the program
Program implementation | 12 months
  Percent of the health facility will implement a minimum standard to program implementation
Maintenance | 24 months
  Percentage of the health facility that will implement a minimum standard to program implementation during the maintenance period

SECONDARY OUTCOMES:
Blood Pressure | 12 months
  Difference in mean systolic and diastolic blood pressure (mmHg) between study arms
Hypertension Diagnosis Awareness | 12 months
  Difference in proportion of patients aware of their HTN diagnosis between study arms
Blood Pressure Control | 12 months
  Difference in proportion of patients with controlled BP (less than 140/90 mmHg) between study arms
Physical activity | 12 months
  Proportion of patients with low physical activity (less than 600 MET-minutes per week) between study arms
Fruits and Vegetables | 12 months
  Proportion of participants with intake of 5 or more servings of fruits and vegetables per day between study arms
Medication | 12 months
  Proportion of participants adherent to hypertension medication between study arms
Affordability | 12 months
  Total incremental costs of care in the study arms
Equity | 12 months
  Household economic impacts in the study arms by measurement of financial and economic costs. Disaggregated analysis, based on gender, ethnicity, and socio-economic status, will be conducted to assess disparities among the study groups
Scalability | 12 months
  Scenario based and sensitivity analysis for scaling up this intervention at the national level
Cost-effectiveness | 12 months
  calculation of incremental cost effectiveness ratios (ICERs) per person per QALY gained
Cost-effectiveness | 12 months
  calculation of incremental cost effectiveness ratios (ICERs) per person per BP control gained
Scalability | 12 months
  Scenario based and sensitivity analysis for scaling up this intervention at the provinical level

CONTACTS AND LOCATIONS:
Overall Officials: Donna Spiegelman, ScD, Principal Investigator — Yale University
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: No